CLINICAL TRIAL: NCT01147302
Title: A Randomized Double-Blind Placebo-Controlled Pilot Study to Evaluate the Safety and Effect of CINRYZE® (C1 Esterase Inhibitor [Human]) for the Treatment of Acute Antibody-Mediated Rejection in Recipients of Donor-Sensitized Kidney Transplants
Brief Title: A Pilot Study to Evaluate the Use of C1 Esterase Inhibitor (Human) in Patients With Acute Antibody-Mediated Rejection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0624-201; 2012-000441-12 (EudraCT Number)
Record Dates: First submitted 2010-06-16; First posted 2010-06-22 (Estimated); Results first posted 2015-07-09 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Graft Rejection
MeSH Terms: interventions — Complement C1 Inhibitor Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- C1 Esterase Inhibitor (Human) (Experimental): Subjects were to receive C1 esterase inhibitor intravenously at a rate of approximately 1 mL per minute as tolerated. Subjects were to receive a total of 7 doses over a 2-week period: an initial IV infusion of 5000 U (not to exceed 100 U/kg) on Day 1, followed by 2500 U (not to exceed 50 U/kg) IV on Days 3, 5, 7, 9, 11, and 13
  Interventions: Biological: C1 Esterase Inhibitor (Human)
- Normal Saline (Placebo Comparator): placebo infused as above
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Placebo
  Arms: Normal Saline
Biological: C1 Esterase Inhibitor (Human)
  Other Names: C1 INH-nf
  Arms: C1 Esterase Inhibitor (Human)

SUMMARY:
The purpose of this research study is to evaluate the safety, effect, and pharmacology of C1 Esterase Inhibitor (human) in kidney transplant patients with acute Antibody-Mediated Rejection (AMR).

ELIGIBILITY:
Inclusion Criteria include:

* ≥18 years of age.
* Weigh ≥50 kg.
* Donor specific antibody identified.

Exclusion Criteria include:

* Any surgical or medical condition that could interfere with the administration of study drug or interpretation of study results.
* History of allergic reaction to C1 Esterase Inhibitor or other blood products.
* Participation in the active dosing phase of any other investigational drug study within 30 days prior to dosing with study drug.
* Pregnancy or lactation.
* Receipt of any experimental agents for AMR within 1 month prior to the first dose of study drug.
* Any infection that causes hemodynamic compromise.
* History of bleeding or clotting abnormality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-08-24 (Actual); Primary Completion 2013-04-19 (Actual); Study Completion 2013-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- United States (4):
  - ViroPharma Investigative Site, Los Angeles, California
  - ViroPharma Investigative Site, Baltimore, Maryland
  - ViroPharma Investigative Site, Minneapolis, Minnesota
  - ViroPharma Investigative Site, Cincinnati, Ohio
- ViroPharma Investigative Site, Heidelberg, Germany

REFERENCES:
- [Derived] Montgomery RA, Orandi BJ, Racusen L, Jackson AM, Garonzik-Wang JM, Shah T, Woodle ES, Sommerer C, Fitts D, Rockich K, Zhang P, Uknis ME. Plasma-Derived C1 Esterase Inhibitor for Acute Antibody-Mediated Rejection Following Kidney Transplantation: Results of a Randomized Double-Blind Placebo-Controlled Pilot Study. Am J Transplant. 2016 Dec;16(12):3468-3478. doi: 10.1111/ajt.13871. Epub 2016 Jun 27. PMID 27184779

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received an intravenous (IV) infusion of normal saline, at a rate of approximately 1 mL per minute as tolerated, 7 times over a 2-week period: an initial infusion on Day 1, followed by infusions on Days 3, 5, 7, 9, 11, and 13.
- CINRYZE: Participants received an intravenous (IV) infusion of human C1 esterase inhibitor (CINRYZE) at a rate of approximately 1 mL per minute as tolerated. Participants received a total of 7 doses over a 2-week period: an initial IV infusion of 5000 U (not to exceed 100 U/kg) on Day 1, followed by 2500 U (not to exceed 50 U/kg) IV on Days 3, 5, 7, 9, 11, and 13.
Period: Overall Study
Arm/Group | Placebo | CINRYZE
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population, defined as all participants who received at least 1 dose (or any portion of a dose) of study drug (CINRYZE or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | CINRYZE | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (13.0) | 48.6 (12.5) | 48.7 (12.4)
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 3 | 4 | 7
  45 to 64 years | 4 | 4 | 8
  65 to 75 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 3 | 4 | 7

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Resolution of The Qualifying Episode of Antibody-Mediated Rejection (AMR)
Description: The "qualifying" renal allograft biopsy was performed as standard of care within 12 months after transplant and prior to screening. The qualifying biopsy was used to establish the diagnosis of AMR and was evaluated for all of the following to obtain baseline assessments: the presence of C4d, and monocyte or neutrophil infiltration around the peritubular capillaries (PTCs) and/or glomeruli. The Central Pathologist provided the following information from the qualifying biopsy in an AMR Scorecard: C4d Score, Glomerulitis Score, Vasculitis Score, Glomerulosclerosis Score, Chronic Glomerulopathy Score, Interstitial Fibrosis Score, and the Chronic Vasculitis Score. The Banff AMR Scoring System was used to summarize these scores. Resolution determination was made based on clinical criteria (improvement of serum creatinine ± decrease of DSA titer, and/or increase in urine output) and histopathology. The first dose of study drug (Day 1) was administered within 72 hours after qualifying biopsy.
Time Frame: 90 days after start of treatment
Population: The Intent-to-Treat Safety (ITT-S) population, defined as participants who received at least 1 dose (or any portion of a dose) of study drug (CINRYZE or placebo).
Measure: Number; unit: participants
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 9 | 9
participants
  Clinical or histopathological resolution, n=9, 9 | 6 | 7
  Resolution based on clinical criteria, n=6, 7 | 3 | 0
  Resolution based on histopathology, n=6, 7 | 4 | 7

2. Primary Outcome: Change From Baseline in Histopathology Endpoints
Description: The protocol-specified Day 20 (post-treatment) biopsy was compared to the qualifying biopsy to assess changes in histopathology for light and immunofluorescence microscopy. The Central Pathologist provided the following categorical information from the qualifying biopsy in an AMR Scorecard: C4d Score (0-100), Margination Score (0-100) Glomerulitis Score (0-100), Vasculitis Score (0-100), Glomerulosclerosis Score (0-100), Chronic Glomerulopathy Score (0-100), Interstitial Fibrosis Score (0-100), and the Chronic Vasculitis Score (0-100), with 0 being absence of abnormal histopathology. The "qualifying" renal allograft biopsy was performed as standard of care (SOC) within 12 months after transplant and prior to screening for this study. The first dose of study drug (Day 1) was administered within 72 hours after qualifying biopsy. A negative change from baseline indicates that histopathology has improved. Endpoint includes subjects with both Qualifying and Day 20 Biopsies.
Time Frame: Within 72 hours prior to first dose of study drug, Day 20
Population: The ITT-S population, defined as participants who received at least 1 dose (or any portion of a dose) of study drug (CINRYZE or placebo).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 9 | 9
scores on a scale
  C4d score | -45.0 (46.9) | -36.1 (33.4)
  Margination score | -6.0 (14.0) | 12.6 (25.9)
  Glomerulitis score | 6.7 (26.6) | 2.7 (13.6)
  Vasculitis score | -3.9 (7.8) | 3.2 (6.4)
  Glomerulosclerosis score | -1.4 (7.8) | -6.3 (7.9)
  Chronic glomerulopathy score | 0.2 (0.7) | 0 (0.0)
  Interstitial fibrosis score | 5.9 (9.8) | 11.6 (20.9)
  Chronic vasculitis score | -1.7 (18.2) | 2.9 (9.0)
Statistical Analysis 1: Comparison: Placebo vs CINRYZE; Analysis of C4d score; Test type: Superiority or Other; p = 0.6498, ANOVA — The p-value for testing the mean for the treatment difference comparison assessed from ANOVA model analysis for CINRYZE versus placebo; Mean treatment difference = 8.89, 95% CI 2-sided [-24.65 to 42.42]
Statistical Analysis 2: Comparison: Placebo vs CINRYZE; Analysis of margination score; Test type: Superiority or Other; p = 0.0768, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean treatment difference = 18.56, 95% CI 2-sided [1.43 to 35.68]
Statistical Analysis 3: Comparison: Placebo vs CINRYZE; Analysis of glomerulitis score; Test type: Superiority or Other; p = 0.6928, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean treatment difference = -4.00, 95% CI 2-sided [-21.36 to 13.36]
Statistical Analysis 4: Comparison: Placebo vs CINRYZE; Analysis of vasculitis score; Test type: Superiority or Other; p = 0.0508, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean treatment difference = 7.11, 95% CI 2-sided [1.23 to 12.99]
Statistical Analysis 5: Comparison: Placebo vs CINRYZE; Analysis of glomerulosclerosis score; Test type: Superiority or Other; p = 0.2042, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean treatment difference = -4.89, 95% CI 2-sided [-11.34 to 1.56]
Statistical Analysis 6: Comparison: Placebo vs CINRYZE; Analysis of chronic glomerulopathy score; Test type: Superiority or Other; p = 0.3322, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean treatment difference = -0.22, 95% CI 2-sided [-0.61 to 0.17]
Statistical Analysis 7: Comparison: Placebo vs CINRYZE; Analysis of interstitial fibrosis score; Test type: Superiority or Other; p = 0.4723, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean treatment difference = 5.67, 95% CI 2-sided [-7.77 to 9.11]
Statistical Analysis 8: Comparison: Placebo vs CINRYZE; Analysis of chronic vasculitis score; Test type: Superiority or Other; p = 0.5103, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean treatment difference = 4.56, 95% CI 2-sided [-7.25 to 16.37]

3. Secondary Outcome: Change From Baseline in Serum Creatinine
Description: Graft function was assessed by measuring serum creatinine. Serum creatinine level was obtained directly from laboratory results. Baseline was the last value collected prior to first dose of study drug. A negative change from baseline indicates that serum creatinine levels have decreased. Values for Day 90 were collected +/= 14 days.
Time Frame: From Day 1 to Days 20 and 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 9 | 9
mg/dL
  Day 20, n=9,9 | -0.2 (0.6) | -0.1 (0.4)
  Day 90, n=9,8 | -0.1 (0.6) | -0.1 (0.4)
Statistical Analysis 1: Comparison: Placebo vs CINRYZE; Analysis of Day 20; Test type: Superiority or Other; p = 0.7591, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean treatment difference = 0.08, 95% CI 2-sided [-0.35 to 0.51]
Statistical Analysis 2: Comparison: Placebo vs CINRYZE; Analysis of Day 90; Test type: Superiority or Other; p = 0.9533, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean treatment difference = -0.01, 95% CI 2-sided [-0.44 to 0.41]

4. Secondary Outcome: Change From Baseline in Creatinine Clearance
Description: Graft function was assessed by measuring creatinine clearance. Creatinine clearance was calculated by the Cockcroft-Gault formula. Baseline was the last value collected prior to first dose of study drug. A positive change from baseline indicates that the clearance rate has increased. Values for Day 90 were collected +/= 14 days.
Time Frame: From Day 1 to Days 20 and 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 9 | 9
mL/min
  Day 20, n=9,9 | 11.4 (24.2) | 12.9 (26.2)
  Day 90, n=9,9 | 3.4 (17.2) | 8.1 (17.7)
Statistical Analysis 1: Comparison: Placebo vs CINRYZE; Analysis of Day 20; Test type: Superiority or Other; p = 0.9046, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean treatment difference = 1.45, 95% CI 2-sided [-19.34 to 22.24]
Statistical Analysis 2: Comparison: Placebo vs CINRYZE; Analysis of Day 90; Test type: Superiority or Other; p = 0.5895, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean treatment difference = 4.68, 95% CI 2-sided [-10.19 to 19.55]

5. Secondary Outcome: Number of Plasmapheresis Sessions
Description: If necessary, rescue therapy included plasmapheresis. Participating centers used plasmapheresis for desensitization, if necessary, prior to transplant and also for the treatment of acute AMR. Plasmapheresis therapy was performed for the qualifying episode of AMR according to standards at the investigational site and at the discretion of the investigator. Sessions include those prior to first dose. If plasmapheresis therapy occurred on the same day as study drug dosing, study drug was administered after completion of the plasmapheresis session.
Time Frame: From Day 1 through Days 20 and 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 9 | 9
sessions
  Day 1 through Day 20, n=9, 9 | 7.4 (5.2) | 9.0 (3.2)
  Day 1 through Day 90, n=7, 6 | 10.4 (7.6) | 10.7 (4.2)
Statistical Analysis 1: Comparison: Placebo vs CINRYZE; Analysis of Day 1 through Day 20; Test type: Superiority or Other; p = 0.4558, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean treatment difference = 1.56, 90% CI 2-sided [-2.00 to 5.11]
Statistical Analysis 2: Comparison: Placebo vs CINRYZE; Analysis of Day 1 through Day 90; Test type: Superiority or Other; p = 0.9470, ANOVA — [p-value comment as in outcome 2, analysis 1]; Mean treatment difference = 0.24, 90% CI 2-sided [-6.05 to 6.52]

6. Secondary Outcome: Number of Participants Who Required Salvage Splenectomy
Description: If necessary, rescue therapy included splenectomy.
Time Frame: From Day 1 to Day 90
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 9 | 9
participants | 0 | 0

7. Secondary Outcome: Number of Deaths
Time Frame: From Day 1 to Day 90
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 9 | 9
participants | 0 | 0

8. Secondary Outcome: Number of Participants With Allograft Failure
Description: Allograft failure was determined by the presence of the following criteria: current renal allograft nephrectomy and/or a clinical determination that the allograft irreversibly and irrevocably ceased functioning.
Time Frame: From the day of enrollment to Day 90
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 9 | 9
participants | 0 | 0

9. Secondary Outcome: Serum Concentrations of C1 Inhibitor (C1 INH) Antigen
Description: Plasma samples were used for the determination of antigenic C1 INH concentrations. Primary pharmacokinetic (PK) parameters were calculated using baseline-corrected concentration-versus-time data following the last dose and noncompartmental techniques, as appropriate. The following PK parameters were calculated: baseline concentration (Cbaseline), maximum concentration (Cmax), average concentration at steady-state (Cav,ss), time to maximum concentration (tmax), minimum concentration (Cmin), area under the concentration-time curve from time zero to last quantifiable concentration at time t (AUC0-t). Blood was collected on Day 13 at the indicated timepoints. If plasmapheresis was performed on a dosing day, blood samples were obtained before plasmapheresis, prior to study drug administration (post-plasmapheresis), and at time points relative to the start of infusion.
Time Frame: Day 13 pre-plasmapheresis (if performed) and pre-dose then 0.5, 2, 24, 48, 96, 168 and 288 (optional) hours post start of infusion
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 9 | 9
g/L
  Unadjusted Cbaseline, n=9, 9 | 0.149 (0.035) | 0.115 (0.041)
  Cmin, n=9, 9 | 0.131 (0.0366) | 0.129 (0.0462)
  Cmax, n=9, 9 | 0.014 (0.020) | 0.081 (0.033)
  Cavg, n=5, 9 | 0.012 (0.014) | 0.052 (0.037)

10. Secondary Outcome: Serum Concentrations of C1 INH Functional Activity
Description: Plasma samples were used for the determination of functional C1 INH concentrations. Primary pharmacokinetic (PK) parameters were calculated using baseline-corrected concentration-versus-time data following the last dose and noncompartmental techniques, as appropriate. The following PK parameters were calculated: baseline concentration (Cbaseline), maximum concentration (Cmax), average concentration at steady-state (Cav,ss), time to maximum concentration (tmax), minimum concentration (Cmin), area under the concentration-time curve from time zero to last quantifiable concentration at time t (AUC0-t). Blood was collected on Day 13 at the indicated timepoints. If plasmapheresis was performed on a dosing day, blood samples were obtained before plasmapheresis, prior to study drug administration (post-plasmapheresis), and at time points relative to the start of infusion.
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units/mL
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 9 | 9
Units/mL
  Unadjusted Cbaseline, n=9, 9 | 1.24 (0.592) | 0.777 (0.301)
  Cmin, n=9, 9 | 1.02 (0.42) | 0.961 (0.441)
  Cmax, n=9, 9 | 0.147 (0.327) | 0.884 (0.457)
  Cavg, n=6, 8 | 0.205 (0.403) | 0.711 (0.513)

11. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of C1 INH
Description: Plasma samples were used for the determination of antigenic and functional C1 INH concentrations. Primary pharmacokinetic (PK) parameters were calculated using baseline-corrected concentration-versus-time data following the last dose and noncompartmental techniques, as appropriate. The following PK parameters were calculated: baseline concentration (Cbaseline), maximum concentration (Cmax), average concentration at steady-state (Cav,ss), time to maximum concentration (tmax), minimum concentration (Cmin), area under the concentration-time curve from time zero to last quantifiable concentration at time t (AUC0-t). Blood was collected on Day 13 at the indicated timepoints. If plasmapheresis was performed on a dosing day, blood samples were obtained before plasmapheresis, prior to study drug administration (post-plasmapheresis), and at time points relative to the start of infusion.
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 9 | 9
hours
  C1 INH antigen, n=5, 9 | 43.2 [0.00 to 44.9] | 0.55 [0.48 to 21.02]
  C1 INH functional activity, n=6, 9 | 4.07 [0.0 to 47] | 3.88 [0.55 to 45]

12. Secondary Outcome: Area Under The Concentration-Time Curve (AUC) of C1 INH Antigen
Description: Plasma samples were used for the determination of antigenic C1 INH parameters. Primary pharmacokinetic (PK) parameters were calculated using baseline-corrected concentration-versus-time data following the last dose and noncompartmental techniques, as appropriate. The following PK parameters were calculated: baseline concentration (Cbaseline), maximum concentration (Cmax), average concentration at steady-state (Cav,ss), time to maximum concentration (tmax), minimum concentration (Cmin), and area under the concentration-time curve from time zero to last quantifiable concentration at time t (AUC0-t). Blood was collected on Day 13 at the indicated timepoints. If plasmapheresis was performed on a dosing day, blood samples were obtained before plasmapheresis, prior to study drug administration (post-plasmapheresis), and at time points relative to the start of infusion.
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g*h/L
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 9 | 9
g*h/L
  AUC0-48hours, n=5, 9 | 0.590 (0.691) | 2.51 (1.79)
  AUClast, n=9, 9 | 2.24 (4.19) | 8.64 (9.50)

13. Secondary Outcome: Area Under The Concentration-Time Curve (AUC) of C1 INH Functional Activity
Description: Plasma samples were used for the determination of functional C1 INH parameters. Primary pharmacokinetic (PK) parameters were calculated using baseline-corrected concentration-versus-time data following the last dose and noncompartmental techniques, as appropriate. The following PK parameters were calculated: baseline concentration (Cbaseline), maximum concentration (Cmax), average concentration at steady-state (Cav,ss), time to maximum concentration (tmax), minimum concentration (Cmin), and area under the concentration-time curve from time zero to last quantifiable concentration at time t (AUC0-t). Blood was collected on Day 13 at the indicated timepoints. If plasmapheresis was performed on a dosing day, blood samples were obtained before plasmapheresis, prior to study drug administration (post-plasmapheresis), and at time points relative to the start of infusion.
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units*h/mL
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 9 | 9
Units*h/mL
  AUC0-48hours, n=6, 8 | 9.82 (19.3) | 34.1 (24.6)
  AUClast, n=9, 9 | 30.8 (50.6) | 113 (86.7)

ADVERSE EVENTS:
Arm/Group | Placebo | CINRYZE
Serious Adverse Events (participants affected / at risk) | 3/9 | 1/9
Other Adverse Events (participants affected / at risk) | 6/9 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | CINRYZE (N=9)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Transplant rejection (Immune system disorders) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | CINRYZE (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Inflammatory pain (General disorders) | 0 | 1
Medical device complication (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 3
Drug hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Transplant rejection (Immune system disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Perinephric collection (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.